CLINICAL TRIAL: NCT05184166
Title: Hospital Management and 1-year Outcome of Patients Aged 70 Years and Older With Severe COVID-19
Acronym: ELDERCOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2021/S03/10
Record Dates: First submitted 2022-01-07; First posted 2022-01-11 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; Elderly Patient
Keywords: COVID-19; ELDERLY PATIENT
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SARS-COV-2 infection can progress to acute respiratory distress syndrome and require hospitalization in the ICU in 5-20% of affected patients. Age is a major risk factor for developing a severe form and for death. ARDS related to SARS-COV-2 has specific features, including the need for long mechanical ventilation and length of stay and the use of corticosteroid therapy. These specificities are responsible for significant morbidity (neuromyopathy, delirium, post-resuscitation syndrome) and mortality during the first wave (46% at 3 months for the population of patients aged 70 years and over). To investigator's knowledge, no study has evaluated the prognosis in the ICU and the long-term functional outcome of elderly people admitted for a severe or critical form of COVID-19 since the major changes in management (dexamethasone, screening for thrombo-embolic complications, use of high-flow oxygen therapy as first-line treatment...).

Investigator therefore propose a 1-year follow-up of a cohort of patients aged 70 and over hospitalised in a conventional service or in intensive care for a severe or critical form of COVID-19. The objectives are to describe the prognosis and functional outcome of hospitalized elderly patients with severe COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 70 years on admission to hospital
* diagnosis of SARS-CoV-2 infection defined by a positive RT-PCR test
* medical or critical care hospitalisation between 1 July 2020 and 31 August 2021
* who experienced severe hypoxaemic acute respiratory failure defined as at least 4L/min of oxygen during hospitalisation

Exclusion Criteria:

* Oxygen therapy < 4L/min during hospitalisation
* Mc Cabe score 3 (chronic disease fatal at 1 year such as stage IV heart failure, ventilated respiratory failure, metastatic cancer, Child C cirrhosis)
* dementia or cognitive disorders before hospitalisation reported in the medical record
* patient GIR 1 to 4 before hospitalisation reported in the medical file or deduced from the description of the lifestyle
* patient with an ADL score < 4 before hospitalisation reported in the medical record or deduced from the description of lifestyle
* patient living in EHPAD before hospitalisation
* non-French speaking patient
* patient under guardianship or curatorship
* refusal to participate in the study for patients surviving 1 year or refusal by a family member or trusted person

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 70 years and over with severe COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Mortality of patients aged 70 years and over 1 year after diagnosis of SAR-COV2 infection | 6 months
  The mortality was evaluated by the proportion of patients aged 70 years and over who died 1 year after diagnosis of SARS-CoV-2 infection who had severe acute respiratory failure defined by at least 4 L/min of oxygen therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France